CLINICAL TRIAL: NCT01647529
Title: Intra-cameral Penetration of Ganciclovir Following Topical Administration of 0.15% Ganciclovir Gel (VIRGAN©) for CMV Anterior Uveitis / Endotheliitis
Brief Title: Topical Administration of 0.15% Ganciclovir Gel for CMV Anterior Uveitis / Endotheliitis
Acronym: Virgan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Samanthila Waduthantri, Clinical Research Fellow, Clinical Associate, Singapore National Eye Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R733/17/2010
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Cytomegalovirus Anterior Segment Infection; Anterior Uveitis; Endotheliitis
Keywords: Cytomegalovirus; uveitis; endotheliitis; ganciclovir
MeSH Terms: conditions — Uveitis, Anterior; Uveitis; Multiple Acyl Coenzyme A Dehydrogenase Deficiency | interventions — Ganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ganciclovir (Experimental): Treatment with topical ganciclovir ointment
  Interventions: Drug: Ganciclovir

INTERVENTIONS:
Drug: Ganciclovir — Treatment with topical ganciclovir ointment

SUMMARY:
Objective of this study is to investigate the intracameral level of ganciclovir following topical application of 0.15% ganciclovir gel (VIRGAN©) for Cytomegalovirus (CMV) anterior uveitis and endothelitis. Thirty patients who are diagnosed with CMV anterior segment infection, either uveitis or endothelitis, who have a positive aqueous real time PCR (RT-PCR) and/or positive tetraplex PCR for CMV and have not had any form of ganciclovir treatment in the past 1 month, will be recruited in the study after taking an informed consent. with active CMV anterior segment infection confirmed by a positive aqueous real time PCR (RT-PCR) and have not had any form of ganciclovir treatment in the past 1 month were recruited in the study. Patients were given 0.15% ganciclovir gel 1cc 5 times a day for 6 weeks. Following 6 weeks of treatment, tears and aqueous samples will be collected. Aqueous will be sent for RT-PCR for CMV status. Ganciclovir drug level in both tears and aqueous will be measured by HPLC method. Clinically, degree of the intraocular inflammation, Intraocular pressure (IOP) and central corneal thickness (CCT) will be recorded at baseline and post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21 and above
* Patients who are diagnosed with anterior uveitis or endotheliitis with a positive aqueous real time PCR (RT-PCR) and/or positive tetraplex PCR for Cytomegalovirus (CMV)
* Patients with relapses and recurrent anterior segment disease that is PCR positive for CMV in aqueous
* Have not been on VIRGAN or any other form of ganciclovir therapy for the past 1 month
* Consent to undergo anterior chamber tap and give aqueous and tear samples for the study
* Able to undergo relevant tests (corneal pachymetry and laser flare cell photometry)
* Able to come for subsequent follow-up visits

Exclusion Criteria:

* CMV anterior uveitis with associated retinitis
* Other causes of hypertensive anterior uveitis / endotheliitis such as HSV, VZV infection
* Patients who have been on any form of (topical, local or systemic) ganciclovir therapy for the past1 month.
* Patients who are allergic to ganciclovir
* Patients who will require systemic or intra-vitreal ganciclovir therapy
* Immunocompromised patients
* Positive for HIV, Hep B and Hep C
* Not keen on participating in the study
* Patients who are incapable, either by law or mental state, of giving consents in their own right.
* Patients who are either unable or unwilling to keep scheduled appointments and adhere to the other aspects of the protocol
* Patients who are pregnant or breastfeeding
* Any other specified reason as determined by the clinical investigator.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Median concentration of ganciclovir in anterior chamber and ocular surface | 6 weeks
  Following 6 weeks of continuous application of Virgan gel 0.15% 1cc 5 times a day, the patient will be reviewed at the clinic within 3 hours following the last application of the gel.

SECONDARY OUTCOMES:
Correlation of intracameral concentration of virgan with the corneal thickness | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Soon P Chee, Principal Investigator — Singapore National Eye Centre; Gemmy Cheung, Study Chair — Singapore National Eye Centre
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore

REFERENCES:
- [Derived] Waduthantri S, Zhou L, Chee SP. Intra-cameral level of ganciclovir gel, 0.15% following topical application for cytomegalovirus anterior segment infection: A pilot study. PLoS One. 2018 Jan 29;13(1):e0191850. doi: 10.1371/journal.pone.0191850. eCollection 2018. PMID 29377953